CLINICAL TRIAL: NCT02039024
Title: Imaging Non-motor Symptoms of Parkinson's Disease by Novel 18F-DTBZ and Florbetapir F-18 PET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, NJI90OKM, Associate Professor, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 100-4356A
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Parkinson's Disease
Keywords: 18F-DTBZ
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18F- DTBZ for Parkinson's Disease (Experimental): This study will compare the amyloid deposition of brain by florbetapir F-18 PET imaging and monoaminergic function by18F- DTBZ PET in 10 NC group, 30 PD group, 30 PDD group, 20 AD group. We will also analyze monoaminergic function by18F- DTBZ PET in 30 PDI group.
  Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping, healthy subjects, PD, PDD, and AD patients will have 4 visits in this study. PDI patients will have 3 visits in this study. Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.
  Interventions: Drug: 18F- DTBZ

INTERVENTIONS:
Drug: 18F- DTBZ — During this study, subjects will receive a single i.v. administration of approximately 370MBq (10 mCi) 18F- DTBZ immediately prior to imaging. The dosage of DTBZ is 10 nmole. The effective dose in human body is about 5.6 mSV.
  During this study, subjects will receive a single i.v. administration of approximately 370MBq (10 mCi) florbetapir F-18 immediately prior to imaging. The dosage of DTBZ is 10 nmole. The effective dose in human body is about 5.6 mSV.
  The proposed dose for this study is based on our phase I study. At the proposed human dose of 10 mCi, the whole body effective dose (ED) will be approximately 680 mrem. The estimated human ED is expected to be comparable to or below the range of other approved brain imaging agents, such as 18F-FDG (Lin 2010).

SUMMARY:
The primary objective of this protocol is to investigate the monoaminergic (dopamine、serotonin、and norepinephrine ) nervous system and amyloid deposition in Parkinson's disease patients with non-motor symptoms (focus on impulse control disorders and dementia) by novel 18F-DTBZ and Florbetapir F-18 PET imaging.

This study will compare the amyloid deposition of brain by florbetapir F-18 PET imaging and monoaminergic function by18F- DTBZ PET in NC group, PD group, PDD group, AD group.

Investigators will also analyze monoaminergic function by18F- DTBZ PET in PDI group.

DETAILED DESCRIPTION:
Study duration is expected to be completed in a period of 3 year. This study will compare the amyloid deposition of brain by florbetapir F-18 PET imaging and monoaminergic function by18F- DTBZ PET in 10 age-matched healthy subjects (NC group), 30 PD patients without dementia/ICD (PD group), 30 PD patients with dementia (PDD group), and 20 patients with dementia (AD group). We will also analyze monoaminergic function by18F- DTBZ PET in 30 PD patients with ICD (PDI group).

Each evaluable subject involved in this study must fulfill all the inclusion and exclusion criteria according the subject grouping, healthy subjects, PD, PDD, and AD patients will have 4 visits in this study ,as one screening visit, one florbetapir F-18 imaging visit, one 18F-DTBZ imaging visit, and one safety evaluation.PDI patients will have 3 visits in this study, as one screening visit, one 18F-DTBZ imaging visit, and one safety evaluation. Safety measurement will be evaluated by medical history, vital signs, physical examinations, laboratory examinations and collecting of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1.10 healthy subjects : i. Male or female subjects, age range 20~80. ii. Subjects have no known neurological or psychiatric disease. However, mild peripheral neuropathies, such as entrapment syndrome or sciatica are allowed.iii. Subjects who provide a written informed consent prior to study entry.

2.30 subjects with a diagnosis of PD : i. Male or female patients, age range 20~80. ii. Patients should be fulfilled "UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria" as "PD". (Appendix I).iii. Patients should not have any clinical evidence of dementia or ICD. iv. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).

3.30 subjects with a diagnosis of PD with dementia : i. Male or female patients, age range 20~80.ii. Patients should be fulfilled the "Movement Disorders Society diagnostic criteria of PDD as "possible" or "probable" PDD (Emre, 2006). (Appendix II) iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).iv. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).

4.20 subjects with a diagnosis of AD : i. Male or female patients, age range 20~80. ii. Patients should be fulfilled the "DSM-IV-TR Diagnostic criteria for Alzheimer's Disease" as AD. (Appendix III).iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).iv. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).

5.30 subjects with a diagnosis of PD with ICD : i. Male or female patients, age range 20~80. ii. Patients should be fulfilled one of the diagnostic criteria or definition in these ICDs: pathological gambling, hypersexuality, compulsive shopping, compulsive eating, punding, and compulsive medication use (Voon, 2009). (Appendix IV).iii. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).iv. Patients who provide a written informed consent prior to study entry. If the patient is incapable of informed consent, the caregiver may consent on behalf of the patient (the patient must still confirm assent).

Exclusion Criteria:

1. Pregnant or becoming pregnant during the study (as documented by pregnancy testing at screening or at any date during the study according to the PI discretion) or current breast feeding.
2. Any subject who has a clinically significant abnormal laboratory values, and/or clinically significant or unstable medical or psychiatric illness.
3. History of drug or alcohol abuse within the last year, or prior prolonged history of abuse.
4. History of intracranial operation, including thalamotomy, pallidotomy, and/or deep brain stimulation.
5. Any documented abnormality in the brain by CT or MRI of brain, which might contribute to the motor function, such as hydrocephalus, multiple infarction and encephalomalacia, will be excluded. Mild cortical atrophy and non-specific white matter changes will be allowed.
6. Any evidence of secondary parkinsonism (multiple infarcts, intoxication, and hydrocephalus, etc) or other neurodegenerative diseases (multiple system atrophy, progressive supranuclear palsy).
7. History of allergy to radioligands that contain 18F isotope.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To compare the amyloid deposition of brain by florbetapir F-18 PET imaging and monoaminergic function by18F- DTBZ PET | 3 years
  To compare the amyloid deposition of brain by florbetapir F-18 PET imaging and monoaminergic function by18F- DTBZ PET in NC group, PD group, PDD group, AD group.
  During this study, subjects will receive a single i.v. administration of approximately 370MBq (10 mCi) florbetapir F-18 immediately prior to imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Hsin Weng, Principal Investigator — Chang Gung Memory Hospital
Locations (1):
- Chang Gung Memory Hospital, Taoyuan District, Taiwan